CLINICAL TRIAL: NCT04273737
Title: Use of Amantadine in Treating Cognitive and Motor Impairments in Adolescents and Adults With Cerebral Palsy
Brief Title: Amantadine in Treating Cognitive & Motor Impairments in Adolescents and Adults With Cerebral Palsy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left institution.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS1907
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; amantadine; cognitive function; gross motor skills; fine motor skills; mood
MeSH Terms: conditions — Cerebral Palsy | interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amantadine (Experimental): Daily regimen of amantadine hydrochloride tablets for 6 weeks: dosing of 5mg/kg divided by two daily doses (max daily dose of 300 mg)
  Interventions: Drug: Amantadine Hydrochloride

INTERVENTIONS:
Drug: Amantadine Hydrochloride — 6-week long daily regimen of amantadine, twice a day, while documenting perceived effects in a diary.
  Other Names: Symmetrel; Symadine; Osmolex ER; Gocovri

SUMMARY:
Cerebral palsy (CP) is a common childhood-onset disability associated with motor and cognitive impairments, however most research is focused on motor outcomes. The aim of this study is to determine the effects of Amantadine, a dopaminergic agonist, on cognitive function in adolescents and adults with CP.

DETAILED DESCRIPTION:
CP is a heterogeneous condition due to injury to the developing brain. It is a condition that is often marked by both cognitive and motor disorders as well as increased prevalence of depression and anxiety. While most studies have focused on improving motor dysfunction, fewer have investigated cognitive impairments associated with CP. Dedicating a study to research the pharmacotherapeutic effect of Amantadine on cognitive function in adolescents and adults with cerebral palsy fills an important gap in development of a potential innovative treatment for cognitive deficits. The investigators hope to determine the effects of Amantadine on cognitive function in adolescents and adults with CP. The investigators will also evaluate secondary goals of improving gross and fine motor skills and mood.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cerebral Palsy

Exclusion Criteria:

* Currently pregnant
* Unstable seizure condition
* Currently taking methadone
* Currently taking other dopamine agonists
* Currently taking anti-psychotic medication
* Previously taken amantadine
* Diagnosed with Chronic Kidney Disease (CKD)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heakyung Kim, MD, Principal Investigator — Columbia Irving Medical Center
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amantadine
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled.
Arm/Group | Amantadine
Number analyzed (Participants) | 11
Age, Customized [Mean (Standard Deviation); unit: years]
  Ages | 24.8 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 11
Cerebral Palsy Diagnosis [Count of Participants; unit: Participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Brief-A Score
Description: The BRIEF-A is a standardized measure that captures views of an adult's executive functions or self-regulation in his or her everyday environment. Both a self-report and an informant report are used. The BRIEF-A includes 75 items within nine non-overlapping theoretically and empirically derived clinical scales: Inhibit, Self-Monitor, Plan/Organize, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and Organization of Materials. All 75 items are rated in terms of frequency on a 3-point scale: 1 (never), 2 (sometimes), 3 (often). Raw scores for each scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Composite scores are calculated and are scored from a range of 75 (better outcome) to 225.
Time Frame: Baseline
Population: Only includes collected data from participants who completed the BRIEF-A at baseline.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Amantadine
Number analyzed (Participants) | 7
T-score | 57.4285 (8.050)

2. Secondary Outcome: Mean PHQ-9 Score
Description: The Patient Health Questionnaire (PHQ-9) is a self-administered, nine-item depression scale of the patient health questionnaire. The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV.
  The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total scores can range from 0 to 27.
  A total score of 0-4 indicates minimal depression severity, 5-9 indicates mild depression severity, 10-14 indicates moderate depression severity, 15-19 indicates moderately severe, 20-27 indicates severe depression severity. Therefore, a high score indicates a worse outcome.
  Outcome measures will be assessing a change in scores pre- and post- prescription of Amantadine.
Time Frame: Baseline
Population: Only includes the collected data from participants who completed the PH-9 at the baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine
Number analyzed (Participants) | 9
score on a scale | 4.667 (4.397)

3. Secondary Outcome: Mean PHQ-9 Score
Description: as for outcome 2
Time Frame: 3 weeks
Population: Only includes the collected data from participants who completed the PH-9 at the 3-week visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine
Number analyzed (Participants) | 7
score on a scale | 3.14 (1.726)

4. Secondary Outcome: Mean PHQ-9 Score
Description: as for outcome 2
Time Frame: 6 weeks
Population: Only includes the collected data from participants who completed the PH-9 at the 6-week visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Amantadine
Number analyzed (Participants) | 7
score on a scale | 6.429 (5.473)

5. Primary Outcome: Mean Brief-A Score
Description: as for outcome 1
Time Frame: 3 weeks
Population: Only includes the collected data from participants who completed the BRIEF-A at the 3-week visit.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Amantadine
Number analyzed (Participants) | 5
T-score | 55.2 (9.431)

6. Primary Outcome: Mean Brief-A Score
Description: as for outcome 1
Time Frame: 6 weeks
Population: Only includes the collected data from participants who completed the BRIEF-A at the 6-week visit.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Amantadine
Number analyzed (Participants) | 5
T-score | 60.2 (10.979)

ADVERSE EVENTS:
Time Frame: Baseline to 6 weeks
Arm/Group | Amantadine
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine (N=11)
Seizure event (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine (N=11)
Increased Muscle Ridigity (Muscle tone) (Musculoskeletal and connective tissue disorders) | 1 (1)
Possible Urinary retention, dizziness, dullness (Gastrointestinal disorders) | 1 (1)
Right Hip pain for 3 days (with collapse due to pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Mania (Nervous system disorders) | 1 (1)
urinary Tract Inflection (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT04273737/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT04273737/ICF_001.pdf